CLINICAL TRIAL: NCT05493839
Title: A Reverification of the Berlin Definition Plateau Criteria in Golmud
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, doctor, Southeast University, China
Other Study IDs: ARDS in Golmud
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Ards
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Plateau Criteria: mild ： 142mmHg < PaO2/ FiO2 ≤ 213 mmHg moderate ： 71mmHg < PaO2/ FiO2 ≤ 142mmHg severe： PaO2/ FiO2 ≤ 71 mmHg
- Berlin Definition: mild ： 200mmHg < PaO2/ FiO2 ≤ 300 mmHg moderate ： 100mmHg < PaO2/ FiO2 ≤ 200mmHg severe： PaO2/ FiO2 ≤ 100 mmHg
- zhang: ARDS：PaO2/FiO2≤100mmHg ALI ：100mmHg<PaO2/FiO2≤150mmHg

SUMMARY:
This study is a single-center retrospective study. According to the Berlin diagnostic standard, ARDS patients admitted to the Department of severe Medicine, Golmud People's Hospital from January 2015 to june 2022 were divided into three groups: mild (142mmHg < PaO2/ FiO2 ≤ 213 mmHg), moderate (71mmHg < PaO2/ FiO2 ≤ 142mmHg) and severe (PaO2/ FiO2 ≤ 71 mmHg). The ICU mortality, 28-day mortality, non-ventilator time in ICU, ICU hospitalization time observed respectively.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of ARDS

Exclusion Criteria:

* length of stay in hospital less than 48h Data missing younger than 18 years or older than 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a single-center retrospective study. According to the Berlin diagnostic standard, ARDS patients admitted to the Department of severe Medicine, Golmud People's Hospital from January 2015 to june 2022 were divided into three groups: mild (142mmHg < PaO2/ FiO2 ≤ 213 mmHg), moderate (71mmHg < PaO2/ FiO2 ≤ 142mmHg) and severe (PaO2/ FiO2 ≤ 71 mmHg).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | up to 24 weeks
  Mortality during treatment in ICU
28-days mortality rate | up to 24 weeks
  28-days mortality rate [ Time Frame: 28 days after discharge ] Mortality at 28 days of hospitalization

SECONDARY OUTCOMES:
Ventilator Free time | up to 24 weeks
  Ventilator Free time in ICU
Ventilator time | up to 24 weeks
  Ventilator time in ICU
Hospital length of stay | up to 24 weeks
  Hospital length of stay in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China